CLINICAL TRIAL: NCT07020871
Title: Correlation of Dry Eye Disease, Problematic Smartphone Use and Sleep Quality in Adolescents and Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, PhD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2024KYPJ090
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease (DED)
Keywords: dry eye disease; problematic smartphone use; sleep quality; bedtime procrastination; adolescents and young adults
MeSH Terms: conditions — Dry Eye Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Investigation Team: 1. After informed consent, adolescents and young adults aged 14-35 years old (including 14,35 years old) are assessed by questionnaires and dry eye related examinations.
  2. The main content is Investigating the relationship among dry eye disease, problematic smartphone use, bedtime procrastination, and sleep quality.

SUMMARY:
The goal of this observational study is to learn about the status quo and relationship of dry eye, problematic smartphone use, bedtime procrastination, and sleep in adolescents and young adults. The main questions it aims to answer are:

* Is there a positive correlation between problematic smartphone use and dry eye?
* Is problematic smartphone use positively correlated with bedtime procrastination?
* Is bedtime procrastination negatively correlated with sleep quality?
* Is there a negative correlation between sleep quality and dry eye?
* Is there a negative correlation between problematic smartphone use and sleep quality?
* Is there a positive correlation between bedtime procrastination and dry eye?
* Do bedtime procrastination and sleep quality serve as mediating factors in the relationship of problematic smartphone use and dry eye? Participants will be asked to complete several questionnaires and dry eye related examinations.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults aged 14 to 35 (including 14,25 years old) ;
* Agree to participate in the studies

Exclusion Criteria:

* Unable to communicate normally;
* With ocular surface diseases other than dry eye and autoimmune diseases;
* Use drugs that may cause damage to the ocular surface, such as anti glaucoma drugs, antidepressants, sex hormones, chemotherapy drugs, etc.;
* With a history of eye trauma or eye surgery;
* With a history of wearing contact lenses within the past month;
* Pregnant and lactating women

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General adolescents and young adults between 14-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 453 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dry eye symptoms | baseline
  Ocular Surface Disease Index scale with 12-item will be used to measure dry eye symptoms. The scale uses Likert 5 comments, with a total score ranging from 0 to 100. And the total score reaching or exceeding 13 points indicates that participants exhibit symptoms of dry eye.
Problematic smartphone use | baseline
  The 10-item Smartphone Addiction Scale Short Version will be used to measure the problematic smartphone use. The scale uses Likert 6 comments, with a total score ranging from 10 to 60. And higher scores indicate more severe problematic smartphone use.
sleep quality | baseline
  The Pittsburgh Sleep Quality Index scale is used to measure participants' sleep quality. The total score ranges from 0 to 21. Higher scores indicate lower quality of sleep.
bedtime procrastination | baseline
  There are 9 items in the Bedtime Procrastination Scale, which is used to measure participants' bedtime procrastination. The scale uses 5-point scale, with a total score ranging from 9 to 45. And higher scores indicate more severe procrastination before sleep.

SECONDARY OUTCOMES:
Perceived level of stress | baseline
  The 14-item Chinese Perceived Stress Scale will be used to measure the perceived level of stress among adolescents and young adults. The scale uses Likert 5 comments, with a total score ranging from 0 to 56. And higher scores indicate a greater pressure that individuals feel in their daily lives.
non-invasive tear film break-up time | baseline
  Non-invasive tear film break-up time is measured by Oculus Keratograph 5M. A cut-off value of less than or equal to 10 s has been reported to be indicative of DED.

OTHER OUTCOMES:
Tear meniscus height | baseline
  The Ocular Keratograph 5M was utilized to measure the tear meniscus height directly beneath three points: the center of the pupil, the nasal corneal limbus, and the temporal corneal limbus. The average of these three measurements was calculated to serve as the final data for tear meniscus height.
Meibomian gland loss | baseline
  The degree of Meibomian gland loss was scored according to the meiboscore (Grade 0: no dropout, Grade 1: dropout of 2/3 of lid area, Grade 2: dropout of 1/3-2/3 of lid area, Grade 3: dropout of >2/3 of lid area).
Lipid layer thickness (LLT) and blinking pattern | baseline
  The LLT and blinking pattern were assessed using LipiView interferometer. The LLT information included the minimum, maximum, and average for 20 seconds. The blinking pattern was obtained by determining the total blinking and partial blinking rates in 20 seconds and then calculating the partial blinking/total blinking ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No